CLINICAL TRIAL: NCT06824701
Title: A Phase 1b Study of Tazemetostat in Combination With Zanubrutinib and Anti-CD20 Monoclonal Antibody in Relapsed or Refractory Indolent B-cell Non-Hodgkin Lymphomas (TARZAN Trial)
Brief Title: Tazemetostat in Combination With Zanubrutinib and Anti-CD20 Monoclonal Antibody in Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Acronym: TARZAN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI183680
Record Dates: First submitted 2025-01-16; First posted 2025-02-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — tazemetostat; zanubrutinib; Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: All Patients (Experimental): The study will investigate the effectiveness of Tazemetostat in combination with Zanubrutinib and anti-CD20 monoclonal antibody
  Interventions: Drug: Tazemetostat; Drug: Zanubrutinib; Drug: Rituximab; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat will be self-administered BID as an oral treatment on a 28-day cycle.
  Other Names: Tazverik
Drug: Zanubrutinib — Zanubrutinib will be self-administered BID as an oral treatment on a 28-day cycle.
  Other Names: Brukinsa
Drug: Rituximab — Rituximab or a biosimilar will be administered intravenously per standard of care.
  Other Names: Ruxience; Rituxan
Drug: Obinutuzumab — Obinutuzumab will be administered intravenously on days 1, 8, 15 of cycle 1 and then day 1 of cycles 2 to 12.
  Other Names: Gazyva

SUMMARY:
The purpose of this clinical trial is to learn if the study drug Tazemetostat combined with Zanubrutinib and anti-CD20 monoclonal antibody is safe and effective in treating patients with relapsed or refractory indolent B-cell non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥ 18 years.
* Eligible histologies include MCL, MZL (including splenic, nodal, and extranodal sub-types), and WM who received at least one line of prior systemic therapy and FL who received at least two prior lines of systemic therapy
* Measurable disease: at least one lesion >1.5 cm in longest diameter or 1 extranodal lesion >1 cm in the longest diameter.

  --Note: For MZL, isolated splenomegaly and involvement of any biopsy proven extranodal site is considered measurable for this study. For MCL, clonal lymphocyte measured by flow cytometry is considered measurable. For WM, serum IgM level >0.5 g/dL is considered measurable.
* Patients must have an indication for treatment.

  * For R/R FL: active disease requiring treatment
  * For R/R MCL: active disease requiring treatment
  * For R/R MZL: active disease requiring treatment
  * For R/R WM: Meeting at least 1 criterion for treatment according to consensus panel criteria from the Seventh International Workshop on Waldenstrom's Macroglobulinemia68

    * Recurrent fever, night sweats, weight loss, fatigue
    * Hyperviscosity
    * Lymphadenopathy which is either symptomatic or bulky (≥ 5 cm in maximum diameter)
    * Symptomatic hepatomegaly and/or splenomegaly
    * Symptomatic organomegaly and/or organ or tissue infiltration
    * Peripheral neuropathy due to WM
    * Symptomatic cryoglobulinemia
    * Cold agglutinin anemia
    * Immune hemolytic anemia and/or thrombocytopenia related to WM
    * Nephropathy related to WM
    * Amyloidosis related to WM
    * Hemoglobin <10 g/dL
    * Platelet count <100,000/mm3
* ECOG Performance Status ≤ 2.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥750 cells/mm3 (≥0.75 x 10^9/L) independent of G-CSF support
    * Platelet count ≥75,000 cells/mm^3 (≥75 x 10^9/L) independent of transfusion support.
  * Hepatic:

    * Total Bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN with document liver involvement and/ or Gilbert's disease.
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN ----Subjects with liver involvement will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
  * Renal:
  * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:
* Adequate coagulation, defined as activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) and prothrombin (PT) or (international normalized ratio (INR) not greater than 1.5 x ULN.
* Life expectancy of >3 months, in the opinion of the investigator
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception and lactation requirements as described in Section 5.3.1 and 5.3.2.
* Subjects must agree to not breastfeed while on treatment or within 1 week of the last dose of tazemetostat or 2 weeks of zanubrutinib.
* Ability to swallow oral tablets
* Patients or their legal representatives must be able to read, understand, and provide informed consent to participate in the trial.
* Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* Time between prior anticancer therapy and first dose of tazemetostat as below:

  * Cytotoxic chemotherapy - At least 21 days
  * Non-cytotoxic chemotherapy (e.g., small molecule inhibitor) - At least 14 days
  * Monoclonal antibody(ies) - At least 28 days
  * Radiotherapy

    * At least 14 days from local site radiation therapy
    * At least 6 weeks from prior radioisotope therapy
    * At least 12 weeks from 50% pelvic or total body irradiation
  * High-dose therapy with autologous hematopoietic cell infusion - At least 60 days
  * CART cell therapy - At least 60 days
  * Moderate CYP3A inhibitors - At least 3 elimination half-lives
  * Moderate CYP3A inducers - At least 14 days
  * Strong CYP3A inducers or inhibitors - At least 14 days ----Note: Must be able to obtain zanubrutinib and anti-CD20 mAb commercially

Exclusion Criteria:

* Prior exposure to tazemetostat or other inhibitor(s) of EZH2
* Any prior history of myeloid malignancies including MDS/AML or MPN
* Any prior history of T-LBL, T-ALL, or B-ALL
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the study drugs
* Major surgery within 4 weeks prior to enrollment
* Known history of bleeding diathesis or active bleeding
* Known history of stroke or intracranial hemorrhage within 6 months of enrollment
* Significant cardiovascular disease defined as:

  * unstable angina or acute coronary syndrome within the past 2 months prior to study enrollment
  * history of myocardial infarction within 3 months prior to study enrollment or documented LVEF by any method of ≤ 40% in the 12 months prior to study enrollment --≥ Grade 3 NYHA functional classification system of heart failure, uncontrolled or symptomatic arrhythmias
* Significant liver disease (>Child Pugh Class A)
* Patients with CNS involvement
* Prolongation of the QT interval corrected for heart rate (QTcF) > 480 msec. QTcF is calculated using Fridericia's Formula (QTcF): QTcF = QT/(RR0.33).

  * Correction of suspected drug induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.
  * Correction for underlying bundle branch block (BBB) allowed. ---Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
* Patients who have tested positive for Human Immunodeficiency Virus (HIV)
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below:

  * Hepatitis B virus (HBV): Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation before enrollment. Patients who are HBV DNA PCR positive will be excluded. Patients with positive anti-HBc and negative HBV DNA should be on prophylactic nucleo(t)side analogue therapy to prevent reactivation with serial HBV DNA PCR monitoring (see the section on "General guidance for hepatic monitoring")
  * Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before enrollment. Patients who are hepatitis C RNA positive will be excluded.
* Known Cytomegalovirus (CMV) infection.
* Evidence of other clinically significant uncontrolled condition(s) including but not limited to, uncontrolled systemic bacterial, viral, fungal, or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the investigator and medical monitor may pose a risk for patient participation. Screening for chronic conditions is not required.
* Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts.
* Active second malignancy unless in remission and with life expectancy > 2 years.
* Patients requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist.
* Receipt of live virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment
* Have a known hypersensitivity to any of the excipients of tazemetostat.
* Subjects taking medications that are known strong CYP3A4 inducers or inhibitors and cannot come off the medication.
* Subjects taking medications that are known moderate CYP3A inducers and cannot come off the medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of tazemetostat in combination with zanubrutinib and anti-CD20 mAb | 2 years
  To determine the MTD of tazemetostat in with zanubrutinib and anti-CD20 mAb. MTD is the highest dose where 0 of the first 3 or 1 of 6 patients had a dose-limiting Toxicity (DLT) during Cycle 1 of tazemetostat treatment.
  This will report the number of patients with DLTs at Dose Level (DL)-1, DL1, and DL2. A DLT is:
  A Grade ≥ 3 non-hematologic toxicity lasting >3 days EXCEPT:
  * Alopecia
  * Grade 3 fatigue, asthenia, anorexia, constipation, nausea, vomiting, or diarrhea not requiring tube feeding, total parenteral nutrition, or hospitalization
  * Grade 3 or 4 tumor lysis syndrome (resolved ≥7 days) or electrolyte abnormalities (resolved to < Grade 2 in <72 hours)
  * Grade 3 alkaline phosphatase, gamma-glutamyl transferase, amylase, or lipase elevation < 72 hours.
  Any of these hematologic toxicities:
  * Grade 4 neutropenia, febrile neutropenia, or thrombocytopenia
  * Grade 5 hematologic toxicity
  Dose delay due to toxicity > 28 days

SECONDARY OUTCOMES:
Overall response rate (ORR) rate at Cycle 7 Day 1 (C7D1) | 8 months
  To evaluate the ORR at C7D1. ORR is the proportion of patients who had a treatment outcome of Partial Response (PR), Very Good Partial Response (VGPR), or Complete Response (CR).
  CR is the absence of serum monoclonal Immunoglobulin M (IgM) protein by immunofixation, normal serum IgM level, resolution of extramedullary disease, and normal bone marrow aspirate and trephine biopsy.
  VGPR is detectable monoclonal IgM protein, ≥90% reduction in serum IgM level, complete resolution of extramedullary disease, and no new signs of active disease.
  PR is detectable Monoclonal IgM protein, ≥50% but < 90% reduction in serum IgM, reduction in extramedullary disease, and no new sign of active disease.
  These are based on the response criteria for Waldenstrom Macroglobulinemia (WM) developed by the International Workshop on WM (IWWM), updated in the sixth IWWM.
  ORR indicates that treatment was effective. This outcome measure will report the proportion of patients who achieve ORR at C7D1.
Very Good Partial Response (VGPR) Rate at Cycle 7 Day 1 (C7D1) | 8 months
  To evaluate the Very Good Partial Response (VGPR) rate at Cycle 7 Day 1 (C7D1). VGPR is a treatment outcome for t B-cell non-Hodgkin lymphomas characterized by detectable monoclonal IgM protein, ≥90% reduction in serum IgM level from baseline, a complete resolution of extramedullary disease (ie, lymphadenopathy/splenomegaly if present at baseline), and no new signs or symptoms of active disease.
  The response assessment will be based on the consensus-based uniform response criteria for Waldenstrom Macroglobulinemia (WM) developed by the International Workshop on Waldenstrom's Macroglobulinemia (IWWM), updated in the sixth IWWM.
  VGPR is used to indicate that the treatment has been highly effective, leading to substantial but not complete remission. This outcome measure will report the proportion of patients who achieve VGPR at C7D1.
Median Duration of Response (DOR) | 7 years
  To evaluate the Duration of Response (DOR) in participants who achieve response. DOR is defined as for patients who achieve response, the time from initial response to the time of death or progression, whichever occurs first. Participants who still respond at their last follow-up will be censored at that time.
  This outcome measure will report the median DOR and corresponding 95% confidence interval.
Median Progression-Free Survival (PFS) | 2 years
  To evaluate median Progression-Free Survival (PFS) from treatment initiation. PFS is defined as the time from treatment initiation to the time of disease progression or death. Patients who are alive and progression-free will be censored at their last follow-up time. Patients who start a subsequent anticancer therapy will be censored at their last follow-up prior to the start of anticancer therapy.
  This outcome measure will report the median PFS with the corresponding 95% confidence interval.
Progression-Free Survival (PFS) at two years after treatment initiation. | 2 years
  To evaluate Progression-Free Survival (PFS) at two years after treatment initiation. PFS is defined as the time from treatment initiation to the time of disease progression or death. Patients who are alive and progression-free will be censored at their last follow-up time. Patients who start a subsequent anticancer therapy will be censored at their last follow-up prior to the start of anticancer therapy.
  This outcome will report the proportion of patients who remain free from disease progression two years after starting treatment.
Median Overall Survival (OS) | 2 years
  To evaluate median overall survival (OS) from treatment initiation. OS is defined as the time from treatment initiation to the time of death, with participants who are alive at their last follow-up time being censored at that time.
  This outcome measure will report the median OS with the corresponding 95% confidence interval.
Overall Survival (OS) at two years after treatment initiation. | 2 years
  To evaluate Overall Survival (OS) at two years after treatment initiation. OS is defined as the time from treatment initiation to the time of death, with participants who are alive at their last follow-up time being censored at that time.
  This outcome will report the proportion of participants who are still alive two years following the start of their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Narendranath Epperla, MD, MS, FACP, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute at University of Uta, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No